CLINICAL TRIAL: NCT02913027
Title: Can We Improve the Comfort of Pelvic Exams?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philadelphia Urosurgical Associates (Other)
Responsible Party: Principal Investigator, Kristene Whitmore, Physician, Philadelphia Urosurgical Associates
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pelvic Exams
Record Dates: First submitted 2016-09-12; First posted 2016-09-23 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational (No Intervention): ARM: Normal Pelvic Exam Exposures: External Exam followed by speculum exam, followed by bimanual exam
- Experimental Pelvic Exam (Active Comparator): Arm: Changing the order of Pelvic Exam Intervention: External exam, Bimanual Exam, Speculum Exam
  Interventions: Other: External Exam; Other: Bimanual Exam; Other: Speculum Exam

INTERVENTIONS:
Other: External Exam — The pelvic exam will be completed in the following order: external, speculum, bimanual exam in the "Standard" group. In the Experimental group the pelvic exam will be done with external exam, bimanual exam, then speculum exam.
  Arms: Experimental Pelvic Exam
Other: Bimanual Exam
  Arms: Experimental Pelvic Exam
Other: Speculum Exam
  Arms: Experimental Pelvic Exam

SUMMARY:
The purpose of this study is to investigate patients self-reported comfort levels during each section of the pelvic exam.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to investigate the sequence in which physicians perform the pelvic exam, describe and compare the self-reported comfort during each section of the pelvic exam and how comfort during the exam relates to quality of life, self-esteem, and sexual function in English speaking females at least 18 years of age in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking, female patients
* Are able to can read and write English
* Are utilizing outpatient services at an OBGYN outpatient office
* Are scheduled for a well-woman exam

Exclusion Criteria:

* Non-English speaking patients
* Patients who cannot read or write
* Those who are pregnant
* Have an active vaginal infection
* Patients who, otherwise, do not require a speculum exam during their appointment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score: A change of 13mm | Within 1 hour of the exam

SECONDARY OUTCOMES:
Wellbeing quality of life score: Range 0-4. | Within 1 hour of the exam
  High wellbeing 2.5-4.0, Low wellbeing 1.5-2.4, and very low wellbeing 0-1.4
Rosenberg Self-Esteem Score: Scale 10-40 | Within 1 hour of the exam
  Higher numbers indicate higher self-esteem
Female Sexual Function Index-19 | Within 1 hour of the exam
  Score of less than 26.55 indicates sexual dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Kristene Whitmore, MD, Principal Investigator — Philadelphia Urosurgical Associates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams AA, Williams M. A guide to performing pelvic speculum exams: a patient-centered approach to reducing iatrogenic effects. Teach Learn Med. 2013;25(4):383-91. doi: 10.1080/10401334.2013.827969. PMID 24112210
- [Result] Committee on Gynecologic Practice. Committee opinion No. 534: well-woman visit. Obstet Gynecol. 2012 Aug;120(2 Pt 1):421-4. doi: 10.1097/AOG.0b013e3182680517. PMID 22825111
- [Result] Daley AM, Cromwell PF. How to perform a pelvic exam for the sexually active adolescent. Nurse Pract. 2002 Sep;27(9):28, 31-2, 34, 37-9, 43; quiz 44-5. doi: 10.1097/00006205-200209000-00006. PMID 12352766
- [Result] Primrose RB. Taking the tension out of pelvic exams. Am J Nurs. 1984 Jan;84(1):72-4. No abstract available. PMID 6559035
- [Result] Bates CK, Carroll N, Potter J. The challenging pelvic examination. J Gen Intern Med. 2011 Jun;26(6):651-7. doi: 10.1007/s11606-010-1610-8. Epub 2011 Jan 12. PMID 21225474
- [Result] Hilden M, Sidenius K, Langhoff-Roos J, Wijma B, Schei B. Women's experiences of the gynecologic examination: factors associated with discomfort. Acta Obstet Gynecol Scand. 2003 Nov;82(11):1030-6. doi: 10.1034/j.1600-0412.2003.00253.x. PMID 14616277
- [Result] Wijma B, Gullberg M, Kjessler B. Attitudes towards pelvic examination in a random sample of Swedish women. Acta Obstet Gynecol Scand. 1998 Apr;77(4):422-8. PMID 9598951
- [Result] Bernet R, Buddeberg C. [Physician-patient relations in gynecology: expectations and experiences of patients]. Gynakol Geburtshilfliche Rundsch. 1994;34(1):43-9. doi: 10.1159/000272333. German. PMID 8019173
- [Result] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Result] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Result] Wiegel M, Meston C, Rosen R. The female sexual function index (FSFI): cross-validation and development of clinical cutoff scores. J Sex Marital Ther. 2005 Jan-Feb;31(1):1-20. doi: 10.1080/00926230590475206. PMID 15841702
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton, NJ: Princeton University Press
- [Derived] Rinko R, Yu I, Bakillah E, Alper L, Delaney C, Su M, Dawson M, Gracely EJ, Whitmore KE. Sequence of Pelvic Examination Affects Patient-Reported Pain. Female Pelvic Med Reconstr Surg. 2018 Mar/Apr;24(2):150-154. doi: 10.1097/SPV.0000000000000515. PMID 29474289